CLINICAL TRIAL: NCT05753098
Title: Effect of Sildenafil Citrate Compared to Estrogen as Adjuvant Therapy on Improvement of Endometrial Thickness and Treatment of Unexplained Infertility
Brief Title: Effect of Sildenafil Citrate Compared to Estrogen as Adjuvant Therapy for Unexplained Infertility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-22022
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Subfertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Estrogen Replacement Therapy; Sildenafil Citrate; Clomiphene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- estrogen therapy in addition to clomiphene citrate (Experimental): received clomiphene citrate 50 mg (Tecnovula®) orally twice daily from the 2nd to 7th day of the cycle and estrogen (Cyclopregnova® 2mg, white tablets, BAYER Schering pharma), one tablet every 12 hour from day 8th till triggering of ovulation.
  Interventions: Drug: estrogen therapy; Drug: Clomiphene Citrate 50mg
- sildenafil in addition to clomiphene citrate (Experimental): received clomiphene citrate 50 mg (Tecnovula®) orally twice daily from the 2nd to 7th day of the cycle as and Sildenafil (Respatio® 20mg film coated tablets for 5 days) from last day of menstruation till reaching optimal size of follicle and endometrial thickness
  Interventions: Drug: Sildenafil; Drug: Clomiphene Citrate 50mg
- clomiphene citrate alone (Other): received clomiphene citrate 50 mg (Tecnovula®) orally twice daily from the 2nd to 7th day of the cycle as in the first and second groups in addition to placebo tablet.
  Interventions: Drug: Clomiphene Citrate 50mg

INTERVENTIONS:
Drug: estrogen therapy — oral estradiol valerate
  Other Names: white tablet of cycloprogynova
  Arms: estrogen therapy in addition to clomiphene citrate
Drug: Sildenafil — PDE5 inhibitor
  Other Names: Respatio
  Arms: sildenafil in addition to clomiphene citrate
Drug: Clomiphene Citrate 50mg — used for ovulation induction
  Other Names: Technovula

SUMMARY:
. This study aimed to determine and compare the effect of vaginal sildenafil citrate and estradiol valerate on endometrial thickness, blood flow and pregnancy rates in infertile women.

DETAILED DESCRIPTION:
The study is a randomized controlled trial that was carried on 148 infertile women with unexplained infertility. Patients were divided into 3 groups. Group 1 included 48 patients who received oral estradiol valerate (Cyclo-Progynova 2mg, from day 8th till triggering of ovulation), another 50 patients in group 2 received oral Sildenafil (Respatio 20mg/12hr film coated tablets for 5 days starting from last day of menstruation till ovulation), while group 3 was the control one who included 50 patients were given ovulation induction with CC 50mg/12hr from 2nd to 7th day of cycle. Every patient underwent a transvaginal ultrasound to determine ovulation, number of follicles, and pregnancy rates. Miscarriage, ectopic pregnancy, and multiple pregnancies were tracked for 3 months, as were any adverse consequences.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 to 40 years
* unexplained infertility (primary or secondary)
* had a regular menstrual cycle;
* patent tubes;
* husbands with normal semen parameters.

Exclusion Criteria:

* hypotension;
* cardiovascular, hepatic, and renal diseases;
* uncontrolled diabetes mellitus;
* anovulatory infertility;
* ovarian cysts;
* pelvic adhesions;
* hyperprolactinemia;
* abnormal thyroid functions;
* multiple uterine fibroids;
* patients on nitrates;
* suspicion of endometriosis and adenomyosis,
* subjects have known to receive any treatment for fertility in the last six months

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
pregnancy rates | at the end of each of 3 cycles (28 days)
  measure B HCG and detect number of cases get pregnant in each cycle 28 days

SECONDARY OUTCOMES:
ovulation | 3 months
  measuring dominant follicle starting from D9 of the cycle till reaching 18-20mm

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Study Director — Clinical Pharmacy Faculty of Pharmacy Beni-Suef University
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No